CLINICAL TRIAL: NCT03533959
Title: Prospective Observational Study for Lesion of Neoatherosclerosis: The Efficacy of Alirocumab for the Neoatherosclerosis Reaction Investigated by Serial Optical Coherence Tomography
Brief Title: To Evaluate the Efficacy of Alirocumab for Neoatherosclerosis by Using OCT, in Comparison With Standard Statin Therapy
Acronym: POLARIS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kobe University (Industry)
Responsible Party: Principal Investigator, Hiromasa Otake, Principal Investigator, Kobe University
Other Study IDs: KobeU-170179
Record Dates: First submitted 2018-05-11; First posted 2018-05-23 (Actual); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Coronary Artery Disease Progression
Keywords: in-stent neoatherosclerosis; alirocumab
MeSH Terms: interventions — alirocumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- alirocumab therapy group: patients with 10mg daily rosuvastatin and alirocumab at least 75mg every 2 weaks
  Interventions: Drug: Alirocumab
- standard statin therapy group: patient with 10mg daily rosuvastatin and never use alirocumab or other PCSK-9 inhibitor

INTERVENTIONS:
Drug: Alirocumab — the administration of Alirocumab at least 75mg every 2 weeks
  Groups: alirocumab therapy group

SUMMARY:
The aim of this study is to evaluate the efficacy of alirocumab for in-stent neoatherosclerosis by using optical coherence tomography, in comparison with standard statin therapy.

DETAILED DESCRIPTION:
The investigators investigate to evaluate the efficacy of alirocumab for in-stent neoatherosclerosis. The investigators enrolled the patient who performed drug eluting stent implantation and detected in-stent neoatherosclerosis by follow up optical coherence tomography, and categorized into two group; the patients with alirocumab and rosuvastatin the investigatorsre categorized alirocumab therapy group, and the patients with rosuvastatin alone were categorized standard statin therapy group.

The investigators compare these two group for outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. The age at the time of consent acquisition is 20 years old or over.
2. OCT Images that can be analyzed are obtained, and neoatherosclerosis existed in drug eluting stent
3. lipid lowering therapy with rosuvastatin 10 mg or rosuvastatin 10 mg and aliclumab is performed.
4. Baseline OCT was scheduled to be revisited within 6 to 12 months, or already performed.
5. Document consent has been obtained from the subject person to this research.

Exclusion Criteria:

1. Patients who have received treatment with PCSK 9 inhibitor in the past
2. Patients whose treatment was interrupted before follow-up catheterization during the observation period
3. Patients underwent LDL apheresis.
4. In the case that the researchers judges it as inappropriate as the object of this research.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with stent implantation who were performed coronary angiography and optical coherence tomography (OCT) follow-up of the coronary arteries were candidate.
  These patients were implanted drug elutingstent including sirolimus-eluting stents (Cypher, Cordis, Miami Lakes, FL, USA), paclitaxel-eluting stents (Taxus, Boston Scientific, Natick, MA, USA), or everolimus-eluting stents (XIENCE V, Abbott Vascular, Santa Clara, CA, USA). The investigators assessed their OCT examination at the follow-up OCT time and patients who were detected NA on OCT findings were eligible for the presence study.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Estimated)
Dates: Start 2017-12-18 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Lipid index change between baseline and 9 month follow-up | Baseline and 9 month follow-up
  Lipid core arc was measured by every 0.2-mm interval throughout segments with neoatherosclerosis (NA) on optical coherence tomography (OCT) findings. The mean lipid core arc was calculated for each lesion. Then, the lipid index was calculated by multiplying the mean lipid core arc by the lipid core longitudinal length.

SECONDARY OUTCOMES:
Macrophage grade change between baseline and 9 month follow-up | Baseline and 9 month follow-up
  Macrophage arc were measured on OCT images with NA every 0.2-mm intervals and divided 4 groups as follows: grade 0, no mac¬rophage; grade 1, localized macrophage accumulation (<30°); grade 2, clus¬tered accumulation ≥30° and <90°; grade 3, clus¬tered accumulation ≥90° and <270°; and grade 4, clustered accumulation ≥270° and <360° . Macrophage grade was evaluated as summation of 0 to 4 grades across all cross section in NA.

CONTACTS AND LOCATIONS:
Overall Officials: Hiromasa Otake, M.D., Ph.D, Study Chair — Kobe University Graduate School of Medicine
Locations (1):
- Kobe University Graduate School of Medicine, Department of Cardiology, Kobe, Hyōgo, Japan

IPD SHARING:
Plan to Share IPD: Undecided